CLINICAL TRIAL: NCT06458127
Title: Tele-Palliative Care Intervention for Patients With Chronic Graft-Versus-Host Disease
Acronym: cGVHDTele-PC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-077
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft-versus-host Disease; Chronic GVHD; cGVHD
Keywords: Chronic graft-versus-host disease; Chronic GVHD; cGVHD; Hematopoietic stem cell transplant; Stem cell transplant; Bone marrow transplant; Telehealth; Telemedicine; Telecare; Palliative care
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-PC Intervention (Experimental): Participants (individuals with moderate to severe chronic Graft-versus-Host Disease) will receive a monthly at home consultation with a specialty palliative care clinician via a video-conference tele-health visit.
  Interventions: Other: Tele-palliative care visit

INTERVENTIONS:
Other: Tele-palliative care visit — Participants will meet with a specialty palliative care clinician for a video-consultation once a month, and complete three tele-PC consultations in total over a three-to-four-month period. They will also complete self-report assessments at baseline and immediately after the last PC intervention visit, approximately 3-4 months after enrolment.

SUMMARY:
This research study is evaluating the feasibility and acceptability of implementing a telehealth palliative care intervention in patients with moderate to severe chronic graft-versus-host disease.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (cGVHD) is a major cause of morbidity among survivors of allogeneic hematopoietic cell transplantation (HCT) patients. Allogeneic HCT is a potentially curative procedure for a variety of hematologic malignancies and involves infusion of donor cells to establish marrow and immune function. Recent advances in risk determination, treatment (i.e., improved safety, use of a variety of donors), prevention of complications, and reduced-toxicity regimens have expanded the eligible patient population, and increased survival of patients who undergo HCT. However, development of cGVHD is a leading complication of allogenic HCT and impacts over 50% of survivors. It develops 3-18 months post-allogeneic HCT and is a main cause of post-HCT morbidity and mortality.

cGVHD is a debilitating immunologic syndrome which attacks different organs in the body, resulting in a wide range of disruptive and unpredictable symptoms. Additionally, side effects of cGVHD include psychological distress with many patients reporting clinical levels of depression and anxiety. Further, patients with cGVHD are also at high risk for late effects, such as skeletal complications, secondary cancers, cardiovascular disease, and thromboembolic events. As a result of this diverse symptom burden, the side effects and psychological distress from illness, and uncertainty of the illness course, patients living with cGVHD experience diminished QOL. Patients with cGVHD struggle to manage their chronic condition, exacerbated with treatment related side effects of physical symptoms, functional limitations, psychological distress, and impaired QOL. Specialty palliative care clinicians have expertise in complex symptom management, facilitate coping with illness and improvement of QOL in cancer patients. Telehealth in various forms has been long studied as an approach to increase access to care, and a care model for management of chronic diseases. Expanding on prior experience with the specialty palliative care model for HCT patients, the investigators aim to develop a telehealth specialty PC model for patients with moderate to severe cGVHD. In this single-arm pilot study, the investigators will test the feasibility and acceptability of a once a month tele-palliative care appointment over the course of 3 months to address the symptom burden, psychological distress and disease uncertainty of cGVHD patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Adult patients (>18 years)
* 2) Have moderate to severe cGVHD based on their oncology clinician assessment as documented in the electronic health record.
* 3) Ability to comprehend and speak English, and to read and respond to questions in English

Please note that this is a proof-of-concept study, and we only include patients who comprehend, read, and respond to questions in English since the study instruments are all available in English. However, as we have done in prior studies, we will expand the population in a future efficacy trial.

Exclusion Criteria:

* 1) Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believe prohibits informed consent or compliance with study procedures
* 2) Patients who have already consulted or are currently consulting palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the tele-palliative care intervention as measured by the proportion of eligible patients who are approached and agree to participate | Week 12
  To calculate the feasibility of the intervention using the proportion of eligible patients who are approached and agree to participate, with 95% confidence interval.
  The intervention will be deemed feasible if at least 60% of patients with moderate to severe cGVHD agree to participate in the study.
Feasibility of the tele-palliative care intervention as measured by the proportion of enrolled participants who complete at least two of the three intervention visits | Week 12
  To calculate the feasibility of the intervention using the proportion of enrolled participants who complete at least two of the three intervention visits, with 95% confidence interval.
  The intervention will be deemed feasible if at least 70% of participants attend at least two of the three intervention visits.

SECONDARY OUTCOMES:
Acceptability of the tele-palliative care intervention as measured by the Client Satisfaction Questionnaire | Week 12
  To calculate the acceptability of the intervention using the the proportion of participants who score >20 on the Client Satisfaction Questionnaire (CSQ-8) with 95% confidence interval.
  Total scores of CSQ-8 range from 8 to 32, with the higher score indicating greater satisfaction. The proposed intervention will be deemed acceptable if at least 60% of participants score >20 on the CSQ-8.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital (MGH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.